CLINICAL TRIAL: NCT01040728
Title: Randomised, Double-blind, Double-dummy, Placebo-controlled, 4-way Cross-over Study to Characterise the 24-hour FEV1-time Profiles of BI 1744 CL 5μg and 10μg (Oral Inhalation, Delivered by the Respimat® Inhaler) and Tiotropium Bromide 18μg (Oral Inhalation, Delivered by the HandiHaler®) After 6 Weeks of Treatment in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Randomized, Double-Blind, 4-way Crossover Study to Evaluate the Efficacy of of 24 Hour Spirometry Profiles of Inhaled BI 1744 CL and Inhaled Tiotropium Bromide in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.40; 2009-014418-86 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; Tiotropium Bromide

ARMS (4):
- Olodaterol (BI1744) Low (Experimental): Low dose inhaled orally once daily from Respimat inhaler
  Interventions: Drug: Olodaterol (BI1744) Low
- Olodaterol (BI1744) High (Experimental): High dose inhaled orally once daily from Respimat inhaler
  Interventions: Drug: Olodaterol (BI1744) High
- Tiotropium 18 mcg (Active Comparator): 18 mcg inhaled once daily from HandiHaler
  Interventions: Drug: Tiotropium 18 mcg
- Placebo (Placebo Comparator): Olodaterol placebo and/or Tiotropium placebo inhaled once daily
  Interventions: Drug: Placebo (for Olodaterol (BI1744)l); Drug: Placebo (for Tiotropium)

INTERVENTIONS:
Drug: Olodaterol (BI1744) Low — Low dose inhaled orally once daily from Respimat inhaler
  Arms: Olodaterol (BI1744) Low
Drug: Olodaterol (BI1744) High — High dose inhaled orally once daily from Respimat inhaler
  Arms: Olodaterol (BI1744) High
Drug: Tiotropium 18 mcg — 18 mcg inhaled once daily from HandiHaler
  Arms: Tiotropium 18 mcg
Drug: Placebo (for Olodaterol (BI1744)l) — Placebo (olodaterol low and high dose) delivered by Respimat
  Arms: Placebo
Drug: Placebo (for Tiotropium) — Placebo (Tiotropium 18 mcg) delivered by HandiHaler
  Arms: Placebo

SUMMARY:
The study is intended to characterize the lung function profile of BI1744 in Chronic Obstructive Pulmonary Disease (COPD) patients where patients will perform pulmonary function tests at regular intervals for 24 hours at the end of a 6 week treatment period. Each patient will receive all four treatments.

ELIGIBILITY:
Inclusion criteria:

* Patients willing to participate with confirmed diagnosis of COPD
* 40 years of age or older
* having a 10 pack year smoking history
* able to perform serial pulmonary function tests
* able to use both a Dry powder inhaler (DPI) and Respimat device

Exclusion criteria:

* Significant other disease
* clinically relevant abnormal hematology, chemistry, or urinalysis
* history of asthma
* diagnosis of thyrotoxicosis
* paroxysmal tachycardia related to beta agonists
* history of MI within 1 year, cardiac arrhythmia, hospitalization for heart failure within 1 year
* active tuberculosis, cystic fibrosis, clinically evident bronchiectasis
* significant alcohol or drug abuse
* pulmonary resection
* taking oral beta adrenergics
* taking unstable oral steroids
* daytime oxygen
* enrolled in rehabilitation program
* enrolled in another study or taking investigational products
* pregnant or nursing women, women of child bearing potential not willing to use two methods of birth control
* those who are not willing to comply with pulmonary medication washouts

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- United States (3):
  - 1222.40.11003 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1222.40.11001 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1222.40.11002 Boehringer Ingelheim Investigational Site, Tampa, Florida
- Germany (3):
  - 1222.40.49401 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.40.49403 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.40.49402 Boehringer Ingelheim Investigational Site, Hanover
- Netherlands (3):
  - 1222.40.31003 Boehringer Ingelheim Investigational Site, Breda
  - 1222.40.31002 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1222.40.31001 Boehringer Ingelheim Investigational Site, Heerlen
- Norway (3):
  - 1222.40.47003 Boehringer Ingelheim Investigational Site, Arendal
  - 1222.40.47002 Boehringer Ingelheim Investigational Site, Drammen
  - 1222.40.47001 Boehringer Ingelheim Investigational Site, Trondheim

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. The duration of each treatment period was 6 weeks with a 3 week washout period between treatments.
Groups:
- Placebo / Tio 18mcg / Olo 10mcg / Olo 5mcg: Patients were administered placebo in the first period, Tiotropium 18 mcg qd in the second period, Olodaterol 10 mcg qd in the third period and Olodaterol 5 mcg qd in the fourth period.
  Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
- Olo 5mcg / Olo 10mcg / Tio 18mcg / Placebo: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 10 mcg qd in the second period, Tiotropium 18 mcg qd in the third period and placebo in the fourth period.
  Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
- Olo 10mcg / Placebo / Olo 5mcg / Tio 18mcg: Patients were administered Olodaterol 10 mcg qd in the first period, placebo in the second period, Olodaterol 5 mcg qd in the third period and Tiotropium 18 mcg qd in the fourth period.
  Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
- Tio 18mcg / Olo 5mcg / Placebo / Olo 10mcg: Patients were administered Tiotropium 18 mcg qd in the first period, Olodaterol 5 mcg qd in the second period, placebo in the third period and Olodaterol 10 mcg qd in the fourth period.
  Olodaterol was administered via the Respimat inhaler, Tiotropium was administered via the HandiHaler.
Period: Overall Study
Arm/Group | Placebo / Tio 18mcg / Olo 10mcg / Olo 5mcg | Olo 5mcg / Olo 10mcg / Tio 18mcg / Placebo | Olo 10mcg / Placebo / Olo 5mcg / Tio 18mcg | Tio 18mcg / Olo 5mcg / Placebo / Olo 10mcg
Started | 31 | 30 | 31 | 30
Completed | 27 | 19 | 30 | 24
Not Completed | 4 | 11 | 1 | 6
Not completed — Adverse Event | 4 | 8 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1
Not completed — Other reasons not listed above | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, double dummy, placebo- and active-controlled, 4 way crossover trial. 122 patients were assigned randomly to one of 4 treatment sequences in which they received each of 4 treatments, two doses (5 microgram (mcg) or 10 mcg) of Olodaterol (Olo) once daily (qd) delivered via the Respimat inhaler or Tiotropium (Tio) 18 mcg once daily (qd) delivered via the HandiHaler or equivalent placebo. The duration of each treatment period was 6 weeks with a 3 week washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 75

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Area Under Curve 0-12 h (AUC 0-12h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit for the first period, just prior to administration of the first morning dose of randomized treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-12h was calculated from 0-12 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to the am dose on the first day of the first treatment period (study baseline) and -30 min (zero time), 30 min, 60 min, 2 hour (h) , 3 h, 4 h, 6 h, 8 h, 10 h, 12 h relative to am dose after six weeks of treatment
Population: Full analysis set (FAS). FAS is defined as all patients with baseline (pre-dose) data and any evaluable post-dosing data for either of the co-primary endpoints. FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler or Aerolizer Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Tio 18 mcg qd: Tiotropium (Tio) 18 mcg qd (morning) delivered by the HandiHaler
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 106 | 112
Liter | -0.008 (0.019) | 0.189 (0.019) | 0.213 (0.019) | 0.213 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using a mixed model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate; Mean Difference (Final Values) = 0.197, 95% CI [0.163 to 0.231], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.221, 95% CI [0.186 to 0.255], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.221, 95% CI [0.187 to 0.255], Standard Error of Mean 0.017 — Tio 18 mcg qd minus Placebo

2. Primary Outcome: FEV1 Area Under Curve 12-24h (AUC 12-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the -1 hour and -10 minute measurements performed in the morning of the first treatment visit for the first period, just prior to administration of the first morning dose of randomized treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 12-24h was calculated from 12-24 hours post-dose using the trapezoidal rule, divided by the observation time (12h) to report in litres.
Time Frame: 1 h and 10 min prior to the am dose on the first day of the first treatment period (study baseline) and 12 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Placebo: Matching Placebo delivered by the Respimat resp. Aerolizer Inhaler.
- Tio 18 mcg qd: Tiotropium 18 mcg qd (morning) delivered by the HandiHaler
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 107 | 112
Liter | -0.059 (0.018) | 0.094 (0.018) | 0.111 (0.018) | 0.105 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.153, 95% CI [0.117 to 0.188], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.170, 95% CI [0.134 to 0.205], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.164, 95% CI [0.128 to 0.199], Standard Error of Mean 0.018 — Tio 18 mcg qd minus Placebo

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-24 h (AUC 0-24h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose at the first randomized treatment visit for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-24h was calculated from 0-24 hours post-dose using the trapezoidal rule, divided by the observation time (24h) to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h, 4 h, 6h, 8h, 10h, 12 h, 22 h, 23 h, and 23 h 50 min relative to am dose after six weeks of treatment
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 107 | 112
Liter | -0.033 (0.019) | 0.142 (0.018) | 0.158 (0.018) | 0.159 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.175, 95% CI [0.141 to 0.208], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.191, 95% CI [0.157 to 0.225], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.192, 95% CI [0.159 to 0.226], Standard Error of Mean 0.017 — Tio 18 mcg qd minus Placebo

4. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response After First Dose of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of the treatment at the first treatment visit for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-3h was calculated from 0-3hours post-dose using the trapezoidal rule, divided by the observation time (3 h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to the am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h , 3 h, relative to the first dose of treatment period
Population: FAS including all patients with evaluable data for this endpoint after first dose of treatment.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Olo 10 mcg qd: Olodaterol 10 mcg qd (morning delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 107 | 113 | 113 | 111
Liter | 0.018 (0.018) | 0.232 (0.017) | 0.256 (0.017) | 0.169 (0.018)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.214, 95% CI [0.181 to 0.248], Standard Error of Mean 0.017 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.238, 95% CI [0.205 to 0.272], Standard Error of Mean 0.017 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.152, 95% CI [0.119 to 0.185], Standard Error of Mean 0.017 — Tio 18 mcg qd minus Placebo

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Area Under Curve 0-3 h (AUC 0-3h) Response After Six Weeks of Treatment
Description: Response was defined as change from baseline. Study baseline FEV1 was defined as the mean of the available pre-dose FEV1 values prior to the first dose of treatment for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FEV1 AUC 0-3h was calculated from 0-3hours post-dose using the trapezoidal rule, divided by the observation time (3 h) to report in litres.
Time Frame: 1 hour (h) prior and 10 minutes (min) prior to the am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h , 3 h, relative to the first dose of treatment after six weeks of treatment
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 106 | 112
Liter | 0.011 (0.020) | 0.225 (0.019) | 0.255 (0.020) | 0.246 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.214, 95% CI [0.178 to 0.251], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.245, 95% CI [0.208 to 0.282], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.235, 95% CI [0.199 to 0.271], Standard Error of Mean 0.019 — Tio 18 mcg qd minus Placebo

6. Secondary Outcome: Peak FEV1 (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of treatment for the first period. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after the first dose of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and first day of dosing
Population: FAS including all patients with evaluable data for this endpoint after first dose of treatment.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 107 | 113 | 113 | 111
Liter | 0.076 (0.019) | 0.313 (0.019) | 0.342 (0.019) | 0.251 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.237, 95% CI [0.201 to 0.273], Standard Error of Mean 0.018 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.266, 95% CI [0.230 to 0.302], Standard Error of Mean 0.018 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.175, 95% CI [0.138 to 0.211], Standard Error of Mean 0.018 — Tio 18 mcg qd minus Placebo

7. Secondary Outcome: Peak FEV1 (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FEV1 was defined as the mean of the available pre-dose peak FEV1 values prior to first dose of treatment for the first period. Peak FEV1 (0-3h) values were obtained within 0 - 3 hours after the last dose after six weeks of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 106 | 112
Liter | 0.082 (0.020) | 0.290 (0.020) | 0.325 (0.020) | 0.325 (0.020)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.208, 95% CI [0.169 to 0.246], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.243, 95% CI [0.205 to 0.282], Standard Error of Mean 0.020 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.244, 95% CI [0.205 to 0.282], Standard Error of Mean 0.019 — Tio 18 mcg qd minus Placebo

8. Secondary Outcome: Trough FEV1 Response
Description: Response was defined as change from baseline. Study baseline trough FEV1 was defined as the mean of the available pre-dose trough FEV1 values prior to first dose of treatment for the first period. Trough values were the mean of values obtained 23h and 23 h 50 min after the last dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 107 | 112
Liter | 0.003 (0.019) | 0.137 (0.019) | 0.146 (0.019) | 0.161 (0.019)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.134, 95% CI [0.097 to 0.171], Standard Error of Mean 0.019 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.143, 95% CI [0.105 to 0.181], Standard Error of Mean 0.019 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.158, 95% CI [0.120 to 0.195], Standard Error of Mean 0.019 — Tio 18 mcg qd minus Placebo

9. Secondary Outcome: Forced Vital Capacity (FVC) Area Under Curve 0-12 Hours (AUC 0-12h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to first dose of treatment for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 0-12h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to the am dose on the first day of the first treatment period (study baseline) and -30 min (zero time), 30 min, 60 min, 2 h, 3 h, 4 h, 6 h, 8 h, 10 h, 12h relative to last dose after six weeks of treatment.
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 106 | 112
Liter | -0.006 (0.035) | 0.324 (0.034) | 0.321 (0.035) | 0.364 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.330, 95% CI [0.276 to 0.384], Standard Error of Mean 0.028 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.326, 95% CI [0.272 to 0.381], Standard Error of Mean 0.028 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.370, 95% CI [0.316 to 0.424], Standard Error of Mean 0.027 — Tio 18 mcg qd minus Placebo

10. Secondary Outcome: FVC Area Under Curve 12-24 Hours (AUC 12-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to first dose of treatment for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 12-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 h and 10 min prior to the am dose on the first day of the first treatment period (study baseline) and 12 h, 22 h, 23 h, and 23 h 50 min relative to last dose after six weeks of treatment
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 107 | 112
Liter | -0.109 (0.036) | 0.169 (0.035) | 0.155 (0.036) | 0.192 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.278, 95% CI [0.214 to 0.342], Standard Error of Mean 0.033 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.264, 95% CI [0.200 to 0.329], Standard Error of Mean 0.033 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.302, 95% CI [0.238 to 0.366], Standard Error of Mean 0.033 — Tio 18 mcg qd minus Placebo

11. Secondary Outcome: FVC Area Under Curve 0-24 Hours (AUC 0-24h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to first dose of treatment for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 0-24h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h, 4 h, 6h, 8h, 10h, 12 h, 22 h, 23 h, and 23 h 50 min relative to last dose after six weeks of treatment
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 107 | 112
Liter | -0.057 (0.036) | 0.247 (0.035) | 0.226 (0.036) | 0.278 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.304, 95% CI [0.244 to 0.363], Standard Error of Mean 0.030 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.283, 95% CI [0.222 to 0.343], Standard Error of Mean 0.031 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.335, 95% CI [0.275 to 0.395], Standard Error of Mean 0.030 — Tio 18 mcg qd minus Placebo

12. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response
Description: Response was defined as change from baseline. Study baseline FVC was defined as the mean of the available pre-dose FVC values prior to the first dose of treatment for the first period. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate. FVC AUC 0-3h was calculated using the trapezoidal rule, divided by the observation time to report in litres.
Time Frame: 1 hour (h) and 10 minutes (min) prior to the am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h relative to first dose of treatment
Population: FAS including all patients with evaluable data for this endpoint after first dose of treatment.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 107 | 113 | 113 | 111
Liter | 0.053 (0.035) | 0.423 (0.034) | 0.419 (0.034) | 0.316 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.370, 95% CI [0.309 to 0.430], Standard Error of Mean 0.031 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.366, 95% CI [0.306 to 0.426], Standard Error of Mean 0.030 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.262, 95% CI [0.202 to 0.322], Standard Error of Mean 0.030 — Tio 18 mcg qd minus Placebo

13. Secondary Outcome: FVC Area Under Curve 0-3 Hours (AUC 0-3h) Response
Description: as for outcome 12
Time Frame: 1 hour (h) and 10 minutes (min) prior to the am dose on the first day of the first treatment period (study baseline) and -30 min, 30 min, 60 min, 2 h, 3 h relative to last dose of treatment after six weeks of treatment
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 106 | 112
Liter | 0.044 (0.035) | 0.388 (0.034) | 0.397 (0.035) | 0.414 (0.034)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.344, 95% CI [0.287 to 0.401], Standard Error of Mean 0.029 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.353, 95% CI [0.296 to 0.411], Standard Error of Mean 0.029 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.370, 95% CI [0.314 to 0.427], Standard Error of Mean 0.029 — Tio 18 mcg qd minus Placebo

14. Secondary Outcome: Peak FVC (0-3h) Response
Description: Response was defined as change from baseline. Study baseline peak FVC was defined as the mean of the available pre-dose peak FVC values prior to first dose of treatment for the first period. Peak FVC (0-3h) was obtained within 0 - 3 hours after the last am dose of study drug after 6 weeks of treatment. Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 106 | 112
Liter | 0.191 (0.037) | 0.526 (0.036) | 0.537 (0.037) | 0.569 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.334, 95% CI [0.272 to 0.396], Standard Error of Mean 0.031 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.346, 95% CI [0.283 to 0.408], Standard Error of Mean 0.032 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.378, 95% CI [0.316 to 0.440], Standard Error of Mean 0.031 — Tio 18 mcg qd minus Placebo

15. Secondary Outcome: Trough FVC Response
Description: Response was defined as change from baseline. Study baseline trough FVC was defined as the mean of the available pre-dose trough FVC values prior to first dose of treatment for the first period. Trough values were the mean of obtained 23 h and 23 h 50 min after the last dose of study drug after six weeks of treatment . Means are adjusted using a mixed effects model with treatment and period as fixed effects and patient as a random effect and study baseline as a continuous covariate.
Time Frame: Study baseline and 6 weeks
Population: FAS including all patients with evaluable data for this endpoint after six weeks.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd | Tio 18 mcg qd
Number analyzed (Participants) | 105 | 115 | 107 | 112
Liter | -0.001 (0.037) | 0.243 (0.036) | 0.215 (0.037) | 0.255 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.244, 95% CI [0.179 to 0.309], Standard Error of Mean 0.033 — Olo 5 mcg qd minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.216, 95% CI [0.150 to 0.282], Standard Error of Mean 0.033 — Olo 10 mcg qd minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Tio 18 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.256, 95% CI [0.191 to 0.321], Standard Error of Mean 0.033 — Tio 18 mcg qd minus Placebo

16. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events related to treatment (cardiac disorders and investigations).
Time Frame: 6 weeks
Population: Treated set.
Measure: Number; unit: participants
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Tiotropium (Tio) 18 mcg qd: Tiotropium (Tio) 18 mcg qd (morning) delivered by the HandiHaler
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Tiotropium (Tio) 18 mcg qd
Number analyzed (Participants) | 109 | 115 | 113 | 113
participants
  Potassium increased | 1 | 0 | 0 | 0
  Atrial fibrillation | 0 | 0 | 1 | 0
  Palpitations | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg | Tiotropium (Tio) 18 mcg qd
Serious Adverse Events (participants affected / at risk) | 5/109 | 3/115 | 8/113 | 2/113
Other Adverse Events (participants affected / at risk) | 8/109 | 14/115 | 6/113 | 4/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=109) | Olo 5 mcg (N=115) | Olo 10 mcg (N=113) | Tiotropium (Tio) 18 mcg qd (N=113)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac ventricular disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=109) | Olo 5 mcg (N=115) | Olo 10 mcg (N=113) | Tiotropium (Tio) 18 mcg qd (N=113)
Nasopharyngitis (Infections and infestations) | 4 | 8 | 4 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication